CLINICAL TRIAL: NCT01103830
Title: Phase I, Randomized, Parallel Group Study to Evaluate the Effect of Multiple Oral Doses of Eurartesim on the QT/QTc Interval Compared to Riamet, Placebo and Moxifloxacin in Healthy Male and Female Volunteers
Brief Title: Safety Study on the Effect of Eurartesim™ on QT/QTc Interval Compared to Riamet in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: sigma-tau i.f.r. S.p.A. (Industry)
Collaborators: Medicines for Malaria Venture (Other)
Responsible Party: Giovanni Valentini MD Head of Clinical Research Unit 1 Medical Department, Sigma Tau ifr SpA
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ST3073-ST3074-DM-09-006
Record Dates: First submitted 2010-04-12; First posted 2010-04-15 (Estimated); Last update posted 2011-06-17 (Estimated); Status verified 2011-06

CONDITIONS: Malaria, Falciparum
Keywords: P. falciparum Malaria, Eurartesim, ACT
MeSH Terms: conditions — Malaria, Falciparum | interventions — artenimol; Artemether; Moxifloxacin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Group 1 (Experimental): 3 or 4 tablets of Eurartesim™, depending of body weight, (3 tablets for subjects weighting less than 75 kg, 4 tablets for subjects weighting 75 kg or more), once daily from Day 1 to Day 3.
  Administration of Eurartesim will be in fed condition following a high-fat/low-Kcal meal.
  Interventions: Drug: Eurartesim™
- Group 2 (Active Comparator): 4 tablets of Riamet® on Day -1 evening, 4 tablets of Riamet® bid (with an interval of 12 ± 0.5 h), in the morning and in the evening of Day 1 and Day 2, 4 tablets of Riamet® in the morning of Day 3.
  Administration of Riamet® will be in fed condition following a high-fat/low-Kcal meal.
  Interventions: Drug: Riamet®
- Group 3 (Other): 3 or 4 tablets of Eurartesim™ placebo, depending of body weight, (3 tablets for subjects weighting less than 75 kg, 4 tablets for subjects weighting 75 kg or more), once daily from Day1 to Day 3.
  Administration will be in the morning, in fed condition, following a high-fat/low-Kcal meal
  1 tablet of Izilox® (400 mg moxifloxacin) in fed condition following a high-fat/low-Kcal meal, on Day 4 morning.
  Interventions: Other: Placebo and finally Moxifloxacin
- Group 4 (Experimental): 3 or 4 tablets of Eurartesim™, depending of body weight, (3 tablets for subjects weighting less than 75 kg, 4 tablets for subjects weighting 75 kg or more), once daily from Day 1 to Day 3.
  Administration of Eurartesim will be in fed condition following a high-fat/high-Kcal meal.
  Interventions: Drug: Eurartesim™
- Group 5 (Experimental): 3 or 4 tablets of Eurartesim™, depending of body weight, (3 tablets for subjects weighting less than 75 kg, 4 tablets for subjects weighting 75 kg or more), once daily from Day 1 to Day 3.
  Administration of Eurartesim will be in fasting condition.
  Interventions: Drug: Eurartesim™
- Group 6 (Other): 3 or 4 tablets of Eurartesim™ placebo, depending of body weight, (3 tablets for subjects weighting less than 75 kg, 4 tablets for subjects weighting 75 kg or more), once daily from Day1 to Day 3.
  Administration will be in the morning, in fasting condition.
  1 tablet of Izilox® (400 mg moxifloxacin) in fed condition following a high-fat/low-Kcal meal, on Day 4 morning.
  Interventions: Other: Placebo and finally Moxifloxacin

INTERVENTIONS:
Drug: Eurartesim™ — 3 or 4 tablets of Eurartesim™ (40mg Dihydroartemisinin and 320 mg Piperaquine phosphate), depending of body weight (3 tablets for subjects weighting less than 75 kg, 4 tablets for subjects weighting 75 kg or more), once daily from Day 1 to Day 3
  Other Names: Dihydroartemisinin and Piperaquine combination therapy
  Arms: Group 1
Drug: Riamet® — 4 tablets of Riamet® (20mg artemether/120mg lumefantrine) on Day -1 evening, 4 tablets of Riamet® bid (with an interval of 12 ± 0.5 h), in the morning and in the evening of Day 1 and Day 2, 4 tablets of Riamet® in the morning of Day 3.
  Other Names: artemether and lumefantrine combination therapy
  Arms: Group 2
Other: Placebo and finally Moxifloxacin — 3 or 4 tablets of Eurartesim™ placebo, depending of body weight, (3 tablets for subjects weighting less than 75 kg, 4 tablets for subjects weighting 75 kg or more), once daily from Day1 to Day 3.
  1 tablet of Izilox® (400 mg moxifloxacin) on Day 4 morning.
  Other Names: moxifloxacin
  Arms: Group 3
Drug: Eurartesim™ — 3 or 4 tablets of Eurartesim™ (40mg Dihydroartemisinin and 320 mg Piperaquine phosphate), depending of body weight (3 tablets for subjects weighting less than 75 kg, 4 tablets for subjects weighting 75 kg or more), once daily from Day 1 to Day 3.
  Other Names: Dihydroartemisinin and Piperaquine combination therapy
  Arms: Group 4
Drug: Eurartesim™ — 3 or 4 tablets of Eurartesim™ (40mg Dihydroartemisinin and 320 mg Piperaquine phosphate), depending of body weight (3 tablets for subjects weighting less than 75 kg, 4 tablets for subjects weighting 75 kg or more), once daily from Day 1 to Day 3.
  Other Names: Dihydroartemisinin and Piperaquine combination therapy
  Arms: Group 5
Other: Placebo and finally Moxifloxacin — 3 or 4 tablets of Eurartesim™ placebo, depending of body weight, (3 tablets for subjects weighting less than 75 kg, 4 tablets for subjects weighting 75 kg or more), once daily from Day1 to Day 3.
  1 tablet of Izilox® (400 mg moxifloxacin)on Day 4 morning.
  Other Names: moxifloxacin
  Arms: Group 6

SUMMARY:
The aim of such a study is to evaluate the impact of a therapeutic dose of Eurartesim™ compared to Riamet®, after multiple dose administration for 3 days in healthy male and female subjects on electrocardiographic parameters.

DETAILED DESCRIPTION:
The fight against malaria, which the WHO reactivated in 1999 with its Roll Back Malaria programme, emphasizes early curative treatment of malaria, particularly in children, in order to decrease mortality and morbidity. Recent estimates confirm a disturbing persistence of endemic malaria with around 515 million cases and 1.0 million deaths per year.The available range of standard antimalarial drugs is narrow. There are only four classes of compounds, probably with different mechanisms of action: 4-aminoquinolines, amino-alcohols, artemisinin derivatives (isolated from a plant, Artemisia annua), and antifolates and drugs related to them.

From a public health perspective, drug resistance is a critical factor that undermines malaria control.Plasmodium falciparum and resistance to chloroquine and sulfadoxine/pyrimethamine is widespread. At present, natural quinine is still effective against P. falciparum everywhere in the world except partially in South-east Asia and South America, where decreased susceptibility is reported. Only the artemisinin derivatives, used for 15 years in Asia and, more recently in Africa, have not generated clinical resistance. Overcoming or reducing resistance requires the adoption of several strategies; central to these is the use of effective chemotherapy for those who need it. In addition, to new molecules, we need to develop and implement strategies to protect drugs against resistance. Resistance to single-drug therapies will inevitably occur. Drug combinations, which have been standard practice for viral and bacterial diseases, are now being adopted for malaria as well. The artemisinin derivatives in combination with standard antimalarials are now being promoted as the best therapeutic option for treating drug-resistant malaria and retarding the development of resistance.

The aim of the present study is to investigate the effect of this new Artemisinin Combination Therapy (ACT) formulation on electrocardiographic parameters. In the literature no relevant QT prolongation associated with Piperaquine treatment has been reported in not-company sponsored trials but no specific TQT trials have been published. On the contrary it has been reported that quinine, quinidine and halofantrine induced a QT prolongation (from slight to severe).

ELIGIBILITY:
Inclusion Criteria:

* Male or female Caucasian subject ≥ 18 and ≤ 50 years;
* Good general health (by medical history and physical examination);
* For male and female subjects of childbearing potential use a double contraception method;
* For female subjects of childbearing potential only: negative plasma pregnancy test at Screening and at admission in the clinical unit;
* Body mass index (BMI) ≥18 and ≤ 27 kg/m2;
* No clinically relevant abnormalities in blood pressure and heart rate;
* No clinically relevant abnormalities in 12-lead ECG results;
* No clinically relevant abnormalities in results of laboratory tests;
* Registered with the French Social Security in agreement with the French law on biomedical experimentation.

Exclusion Criteria:

* A predictable poor compliance or inability to communicate well with the Investigator;
* Unsuitable veins for repeated venipuncture.
* Evidence of clinically relevant cardiovascular, renal, hepatic, hematological, gastrointestinal, pulmonary, metabolic-endocrine, neurological, urogenital or psychiatric diseases as judged by the Investigator;
* A history of additional risk factors for Torsades des Pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome);
* The use of concomitant medications that prolong the QT/QTc interval;
* Any condition requiring regular concomitant medication, including herbal products and over-the-counter (OTC) medication or predicted need of any concomitant medication during the study;
* Evidence of any clinically significant acute or chronic disease, including known or suspected HIV, hepatitis B virus (HBV) and HCV infection;
* History of relevant clinical allergic reactions of any origin;
* Known hypersensitivity to any of the test materials or related compounds;
* Intake of any medication (except paracetamol, hormonal contraceptives and hormone replacement therapy for postmenopausal women), including OTC medications and herbal products that could affect the outcome of the study, within 2 weeks prior to the first drug administration or less than 5 times the t1/2 of that drug, whichever is the longer;
* Drug abuse;
* Current use of nicotine containing products and the inability to stop using nicotine containing products during confinement in the clinical centre.
* Use of caffeine containing beverages exceeding 500 mg caffeine/day and the inability to refrain from the use of caffeine containing beverages during confinement in the clinical centre;
* Intake of any food or any beverage containing grapefruit or grapefruit juice, orange or pomelo juice within 48 h prior to the first dosing and the inability to stop such intake during the study;
* Blood donation or loss of significant amount of blood within three months prior to the first dosing;
* Positive drug screen;
* Positive serology to HIV (HIV1 and HIV2) and/or HCV antibodies, and/or hepatitis B surface antigen (HBsAG);
* Any other condition that in the opinion of the Investigator would interfere with the evaluation of the results or constitute a health risk for the subject;
* Participation in a drug study within 3 months prior to the first dosing.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 287 (Actual)
Dates: Start 2010-02; Primary Completion 2010-08 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
QTcF interval (Fridericia's correction QT interval) | before study drugs administration, during the 24 hrs post first and third dose and during follow-up
  Group 1,4 and 5 (Day -1: pre-dose, each hour till 13h post-dose. Day 1: pre-dose, 1, 2, 3, 4, 5, and 6 h post-dose. Day 3: pre-dose, each hour till 13h post-dose and then 24h).
  Group 2 (Day -2: pre-dose, each hour till 13h post-dose and then 24h. Day 3: pre-dose, each hour till 13h post-dose and then 24h).
  Group 3 and 6 (Day -1: pre-dose, each hour till 13h post-dose. Day 1: pre-dose, 1, 2, 3, 4, 6, 8, 12 and 24h post-dose. Day 3: pre-dose, pre-dose, each hour till 13h post-dose. Day 4: pre-dose, 1, 2, 3, 4, 6, 8, 12 and 24h post-dose).

SECONDARY OUTCOMES:
Effect of Eurartesim™ administered in different food conditions, on ECG parameters | before study drugs administration, during the 24 hrs post first and last dose and during follow-up
  To evaluate the impact of a therapeutic dose of Eurartesim™ under different food intake conditions on the cardiac activity, as expressed by ECG parameters.
Effect of food on bioavailability of Eurartesim™ | during the 24 hrs post first and last dose
  To evaluate the impact of high-fat/high-Kcal or high-fat/low-Kcal meals on the overall relative bioavailability of Eurartesim™ in respect to no food.
To evaluate differences in PK and ECG profiles according to posology scheme | during the 24 hrs post first and last dose
  To compare, within the Eurartesim™ groups, the PK profiles and the QT intervals of subjects with a body weight below or equal and above 75kg
relationship within the Pk parameters of active substances and ECG parameters | during the 24 hrs post first and last dose
  To evaluate the relationship between the PK parameters of Dihydroartemisinin and Piperaquine and the ECG parameters
to asses general safety and tolerability of Eurartesim™ | during the treatment and follow-up period
  To assess the safety and tolerability of Eurartesim™ under different food intake conditions in healthy subjects

CONTACTS AND LOCATIONS:
Overall Officials: Lionel Hovsepian, MD, Principal Investigator — SGS Aster S.A.S.
Locations (1):
- SGS aster s.a.s, Paris, France

REFERENCES:
- [Derived] Funck-Brentano C, Bacchieri A, Valentini G, Pace S, Tommasini S, Voiriot P, Ubben D, Duparc S, Evene E, Felices M, Corsi M. Effects of Dihydroartemisinin-Piperaquine Phosphate and Artemether-Lumefantrine on QTc Interval Prolongation. Sci Rep. 2019 Jan 28;9(1):777. doi: 10.1038/s41598-018-37112-6. PMID 30692558